CLINICAL TRIAL: NCT02772055
Title: A Multicentre, Randomised, Single Blinded, Parallel-group Study of Moxa Smoke Effect in Moxibustion Treating Knee Osteoarthritis
Brief Title: Efficacy of Moxibustion Therapy With or Without Smoke for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015CB554504-02
Record Dates: First submitted 2016-05-10; First posted 2016-05-13 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Pain
Keywords: Moxa smoke; Moxibustion; Knee osteoarthritis
MeSH Terms: conditions — Pain; Osteoarthritis, Knee | interventions — Moxibustion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- moxibustion group (Experimental): Conventional moxibustion treatment for knee osteoarthritis participants.12 sessions of moxibustion treatment over a period of 4 weeks, 3 sessions per week.Each session will last 30 minutes.
  Interventions: Other: Moxibustion
- smoke-free moxibustion group (Experimental): Conventional moxibustion treatment for knee osteoarthritis participants and have a purification device at the top of the moxibustion to remove the moxa smoke.12 sessions of moxibustion treatment over a period of 4 weeks, 3 sessions per week.Each session will last 30 minutes.
  Interventions: Other: Moxibustion; Other: Moxa smoke purification device

INTERVENTIONS:
Other: Moxibustion — Moxibustion at three acupuncture point(EX-LE04,ST35,ST36).12 sessions of moxibustion treatment over a period of 4 weeks, 3 sessions per week.Each session will last 30 minutes.
Other: Moxa smoke purification device — Investigators place a purification device(Shenzhen Conyson Electronic Technology Co, Ltd,C200 moxa smoke purification device,Shenzhen,China) at the top of the moxibustion to remove the moxa smoke.
  Arms: smoke-free moxibustion group

SUMMARY:
This is a multicentre, randomised, single blinded, parallel-group design clinical trial to assess the effect of moxa smoke in the treatment using moxibustion for Knee Osteoarthritis.

DETAILED DESCRIPTION:
Aim: To assess the effect of moxa smoke in the treatment using moxibustion for knee osteoarthritis.

Design: This is a multicentre, randomised, single blinded, parallel-group design clinical trial. 138 eligible participants will be randomly allocated into 2 groups (moxibustion group or smoke-free moxibustion group) with a 1:1 allocation ratio, and receive 12 sessions of moxibustion treatment over a period of 4 weeks, three sessions per week. Each session will last 30 minutes. The whole study period is 13 weeks, with a 1 week run in period, 4 week treatment phase, and 8 week follow-up phase.The participants will receive moxibustion treatment at three acupoints (EX-LE04,ST35,ST36). In moxa-free smoke moxibustion group, investigators place a purification device(Shenzhen Conyson Electronic Technology Co, Ltd,C200 moxa smoke purification device,Shenzhen,China) at the top of the moxibustion to remove the moxa smoke. The primary measurement outcomes are the mean change in the global scale value of the Western Ontario and McMaster Universities Osteoarthritis Index(WOMAC) pain and function scores from baseline to 4 weeks. The secondary outcomes are the Visual Analogue Scale (VAS) and the patient global assessment. Investigators will assess participants at the second visit (before starting moxibustion treatment) and at the 2, 4, 8, and 12 week respectively after the baseline.

ELIGIBILITY:
Inclusion Criteria:

Participants meeting the following criteria will be included:

1. aged between 40 and 75 years
2. diagnosed with knee osteoarthritis formulated by the American College of Rheumatology (ACR).
3. the average severity of knee pain not more than 7 points on a visual analogue scale for most days during the past month
4. agree not have the paregoric during the whole treatment phase
5. willingness to participate in a randomized study and to sign the informed consent form.

Exclusion Criteria:

Participants will be excluded if they have these experiences:

1. inflammatory diseases, including rheumatoid arthritis, cancer, traumatic injury that might be related to the current knee pai
2. autoimmune disease, uncontrolled hypertension
3. diabetes mellitus requiring insulin injection
4. life-threatening cardiovascular or neurological events within the past year
5. chronic respiratory disease,a haemorrhagic disorder
6. alcohol or drug addiction
7. an active infectious disease including tuberculosis
8. a significant knee joint deformity
9. knee replacement surgery for the affected knee
10. knee arthroscopy within the past year
11. steroid injection in the knee joints within the past 3 months
12. injections in the knee joints or joint fluid injection within the past 6 months
13. accept acupuncture, moxibustion, cupping, or herbal medicine within the past 4 weeks

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in the global scale value of the Western Ontario and McMaster Osteoarthritis Index(WOMAC) score | 4 weeks from baseline

SECONDARY OUTCOMES:
Change in the WOMAC subscales (pain, stiffness, and function) | at baseline(0 week), 2 weeks, 4weeks, 8 weeks and 12 weeks later after allocation
Mean change in Visual Analogue Scale for the pain intensity | Assessing participants at baseline(0 week), 2 weeks, 4weeks, 8 weeks and 12 weeks later after allocation
Change of Patient global assessment score | at 2 weeks, 4weeks, 8 weeks and 12 weeks later after allocation

CONTACTS AND LOCATIONS:
Overall Officials: Yu Shuguang, Professor, Principal Investigator — Chengdu University of Traditional Chinese Medicine
Locations (1):
- Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo L, Liao M, Peng JX, Ma Q, Zhou JY, Zhu LL, Wang X, Chen SS, Yin HY, Wu QF, Zhang CS, Lv P, Tang Y, Yu SG. Comparison of the Efficacy between Conventional Moxibustion and Smoke-Free Moxibustion on Knee Osteoarthritis: A Randomized Controlled Trial. Evid Based Complement Alternat Med. 2019 Mar 14;2019:1291947. doi: 10.1155/2019/1291947. eCollection 2019. PMID 31001350
- [Derived] Zhu LL, Zhou JY, Luo L, Wang X, Peng JX, Chen SS, Yin HY, Wu QF, Zhang CS, Lv P, Tang Y, Yu SG. Comparison of the efficacy between conventional moxibustion and smoke-free moxibustion on knee osteoarthritis: study protocol of a randomized controlled trial. Trials. 2017 Apr 24;18(1):188. doi: 10.1186/s13063-017-1846-2. PMID 28438185